CLINICAL TRIAL: NCT06039683
Title: A Multicountry, Multicentre, Non-interventional, Retrospective Study to Determine Real-world Treatment Patterns and Associated Outcomes After First Line Osimertinib in Patients With Advanced and Metastatic NSCLC EGFRm in the GCC Region
Acronym: TREASURE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00045
Record Dates: First submitted 2023-09-06; First posted 2023-09-15 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
A Multicountry, Multicenter, Non-interventional, Retrospective Study to determine Real-world treatment patterns and associated outcomes after FIRST LINE Osimertinib in patients with advanced and Metastatic NSCLC harboring EGFR-activating mutations in the GCC Region

DETAILED DESCRIPTION:
Osimertinib has demonstrated superior PFS compared to firstgeneration EGFR-TKIs (erlotinib and gefitinib) in the first line setting in clinical trials. There remains a need to consider clinical outcomes in the real-world setting and determine the characteristics of long-term survivors in the real world. It will also be important to determine the subsequent treatment pathways of patients who progress on treatment with Osimertinib

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, all the following inclusion criteria must be fulfilled:

1. Patients with Stage IIIB-IV NSCLC using either AJCC 7th or 8th edition with EGFR mutation.
2. Age 18 or older at index date (specific age may vary according to country-specific guidelines)
3. Treated in the first line with Osimertinib from (April 1st, 2018, until December 31st, 2021).
4. Medical records available at the participating site reflect at least 9 months of follow-up from the index date (unless the patient died within the first 9 months of diagnosis).

Note: specific databases may have additional inclusion criteria which will be detailed in country-specific protocol adaptations and statistical analysis plans (SAPs).

Exclusion Criteria:

Subjects are not eligible for this study if they fulfil any of the following exclusion criteria:

1. Failure to meet one or more of the inclusion criteria.
2. Patients who received curative CRT within 3 months and/or any first-line systemic anti-cancer therapies (SACT) for advanced/metastatic NSCLC for >28 days prior to Osimertinib start.
3. Patients who have prior exposure of I/O therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. 18 years or older patients had pathological/molecular confirmed advanced/metastatic EGFRm NSCLC (including both sensitized and uncommon mutations), with or without previous adjuvant/neoadjuvant chemotherapy, initiating first-line Osimertinib treatment between 1st April 2018 till December 31st, 2021.
  2. Patients who are treated with short doses of chemotherapy or any other targeted therapy for up to 28 days before Osimertinib initiation will still be considered "firstline Osimertinib patients."
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
To describe treatments and sequencing after treatment with first line Osimertinib. | 1st April 2018 till December 31st, 2021.
  Treatments and sequencing after treatment with first line Osimertinib - data on all subsequent lines of treatment, duration and dose changes will be collected until death or last contact or interim data cut-off/end of study period along with disease progression and outcome on the respective line of treatment
To describe real world time to the next treatment or death (rwTTNTD). | 1st April 2018 till December 31st, 2021.
  rwTTNTD, defined as the time in days from and inclusive of the index date until the start date of the next systemic therapy line or death from any cause (in absence of next systemic therapy line). Patients who do not receive a subsequent systemic therapy line or die during the study observation period will have TTNTD right censored at the earliest date of last contact or interim data cut-off date/end of the study period.

CONTACTS AND LOCATIONS:
Locations (7):
- Research Site, Kuwait City, Kuwait
- Research Site, Doha, Qatar
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Al Ain City

REFERENCES:
- See also: Redacted CSR-Synopsis_version1.0 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161R00045&attachmentIdentifier=6a15f98c-0dec-4488-ac6e-f72bb83829dc&fileName=Treasure_study_-Redacted_CSR-Synopsis_version1.0.pdf&versionIdentifier=